CLINICAL TRIAL: NCT05857566
Title: A Randomized, Open-Label Study of the Effect of RDX-002 on Postprandial Triglycerides in Subjects Treated With the Atypical Antipsychotic Drug, Olanzapine
Brief Title: Effect of RDX-002 on Postprandial Triglycerides in Subjects Treated With Olanzapine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Response Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDX-002-22-09
Record Dates: First submitted 2023-04-28; First posted 2023-05-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Drug-induced Weight Gain

STUDY DESIGN:
Intervention Model Description: Phase 1b, randomized, open-label, parallel group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RDX-002 (Experimental): 50 mg oral tablet; 200 mg BID for 7 days
  Interventions: Drug: RDX-002
- Olanzapine (Other): 10 mg oral tablet; 10 mg QD for 14 days
  Interventions: Drug: RDX-002

INTERVENTIONS:
Drug: RDX-002 — A potent, selective, and gut-specific microsomal triglyceride transfer protein (MTP) inhibitor.

SUMMARY:
This Phase 1b Study RDX-002-22-09 has been planned to evaluate the effect of RDX-002 on postprandial triglycerides and ApoB48 levels in normal healthy subjects treated with the atypical antipsychotic drug, olanzapine.

DETAILED DESCRIPTION:
This Phase 1b Study RDX-002-22-09 has been planned to evaluate the effect of RDX-002 on postprandial triglycerides and ApoB48 levels in normal healthy subjects treated with the atypical antipsychotic drug, olanzapine. It is a randomized, open-label, parallel group study that will be conducted at a single study site in the US. Normal, healthy subjects aged 18-50 years and with a body mass index (BMI) of 18-27.5 kg/m2 will be eligible for screening. Screening (Day -28) will begin approximately 28 days prior to Baseline (Day 1). Subjects will be admitted to the clinical research unit (CRU) on the morning of Day -1 and will remain in the CRU until discharge on Day 16.

ELIGIBILITY:
Inclusion Criteria:

* A glycated hemoglobin (HbA1c) level of <5.7% at Screening
* A 12-lead electrocardiogram (ECG) at Screening which, in the opinion of the Investigator, had no abnormalities that compromised safety in this study
* Hematology, clinical chemistry and urinalysis at Screening, the results of which fall within normal parameter ranges and/or are deemed clinically acceptable by the Investigator Exclusion Criteria
* Males and nonpregnant, nonlactating females

Exclusion Criteria:

* Any prior use of or contraindication to atypical antipsychotics
* Concomitant use of drugs known to impact the PK of olanzapine
* Type 1 or Type 2 diabetes
* Recent CV event
* Uncontrolled hypertension
* Fasting triglycerides ≥400 mg/dL
* Fasting glucose ≥100 mg/dL
* Any condition that impacts the absorption of dietary fats
* Significant gastrointestinal disorders
* Gall bladder disease
* Uncontrolled hypothyroidism
* Liver disease or dysfunction
* Renal disease or dysfunction
* Gastrointestinal conditions
* Hematologic disorders
* Active malignancy
* Psychiatric disorder
* History of drug or alcohol abuse
* Pregnant, breastfeeding, or intending to become pregnant
* Use of weight loss products
* Blood donation or loss within 30 days prior to Screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Triglyceride and apolipoprotein B48 (ApoB48) | 7 days
  Efficacy of treatment with RDX-002 on postprandial triglyceride levels and apolipoprotein B48 (ApoB48) levels in normal healthy volunteers treated with 10 mg olanzapine.

SECONDARY OUTCOMES:
Triglyceride Level | 7 days
  Evaluate the effect of treatment with 10 mg olanzapine on postprandial triglyceride levels and ApoB48 levels in normal healthy volunteers
Cmax | 7 days
  Assess the effect of RDX-002 dosing on the steady-state pharmacokinetics (PK) of olanzapine
Fasting Lipids | 7 days
  Assess the effects of olanzapine and olanzapine with RDX-002 on fasting lipids
AUC | 7 days
  Assess the effect of RDX-002 dosing on the steady-state pharmacokinetics (PK) of olanzapine
t1/2 | 7 days
  Assess the effect of RDX-002 dosing on the steady-state pharmacokinetics (PK) of olanzapine

CONTACTS AND LOCATIONS:
Overall Officials: Tricia Stamp, PhD, PA-C, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No sharing of IPD with other researchers.